CLINICAL TRIAL: NCT00625833
Title: A Randomized, Double-Blind Placebo Controlled Trial Of [S,S]-Reboxetine In Patients With Chronic Painful Diabetic Peripheral Neuropathy.
Brief Title: A Trial Of [S,S]-Reboxetine In Patients With Chronic Painful Diabetic Peripheral Neuropathy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for futility following the planned interim analysis.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061037
Record Dates: First submitted 2008-02-14; First posted 2008-02-28 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — O-methyl reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: [S,S]-Reboxetine

INTERVENTIONS:
Drug: Placebo — Oral tablet once a day dosing for 10 weeks.
  Arms: Placebo
Drug: [S,S]-Reboxetine — Oral tablet once a day dosing for 10 weeks.
  Arms: 2

SUMMARY:
This is a trial to investigate the effectiveness and safety of [S,S]-Reboxetine in relieving chronic peripheral pain suffered by patients with diabetes. Some evidence for the effectiveness of [S,S]- Reboxetine in relieving chronic pain has been seen in 3 completed trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race at least 18 years of age
* Diagnosis of painful, distal, symmetrical, sensory-motor polyneuropathy, which is due to diabetes, for at least 1 year
* Patients at Visit 1 must have a score ≥40 mm on the Pain Visual Analogue Scale

Exclusion Criteria:

* Patients with significant hepatic impairment
* Neurological disorders unrelated to diabetic neuropathy that may confuse the assessment of neuropathic pain
* Any pain or other condition that may confound assessment or self-evaluation of the pain due to diabetic neuropathy
* Amputations other than toes
* A current or recent diagnosis (past 6 months) or episode of major depressive disorder and/or uncontrolled depression
* History of transient ischemic attack or stroke
* Myocardial infarction or unstable angina within the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly average pain score | 8 weeks

SECONDARY OUTCOMES:
Responder rates (patients with a 30% reduction from baseline in weekly average pain score and patients with a 50% reduction from baseline in weekly average pain score) | 8 weeks
Change from baseline in weekly average sleep interference scale | 8 weeks
Change from baseline in the total score and each dimension of the Neuropathic Pain Symptom Inventory | 8 weeks
Modified Brief Pain Inventory-Short Form | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (27):
  - Pfizer Investigational Site, Anniston, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mission Viejo, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Winter Haven, Florida
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Tupelo, Mississippi
  - Pfizer Investigational Site, Marionville, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Hamilton, New Jersey
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Myrtle Beach, South Carolina
  - Pfizer Investigational Site, Bartlett, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Czechia (4):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Zlín
- Finland (4):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kokkola
  - Pfizer Investigational Site, Lahti
  - Pfizer Investigational Site, Lohja
- Netherlands (3):
  - Pfizer Investigational Site, Almere Stad
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Venlo
- South Africa (7):
  - Pfizer Investigational Site, Worcester, Cape Town
  - Pfizer Investigational Site, Bloemfontein, Free State
  - Pfizer Investigational Site, Ennerdale, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, KwaDukuza, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town
- Spain (6):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Santiago de Compostela, LA Coruña
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Pontevedra
  - Pfizer Investigational Site, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061037&StudyName=A%20Trial%20Of%20%5BS%2CS%5D-Reboxetine%20In%20Patients%20With%20Chronic%20Painful%20Diabetic%20Peripheral%20Neuropathy.